CLINICAL TRIAL: NCT01267877
Title: Patient Perception of Mammogram Guidelines
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: OBGYN13730
Record Dates: First submitted 2010-12-22; First posted 2010-12-29 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Attitude; Practice Guideline; Breast Cancer
Keywords: U.S. Preventive Services Task Force; Patient attitude; Mammogram; Guideline
MeSH Terms: conditions — Behavior; Breast Neoplasms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Guideline unfavorable article (Active Comparator)
  Interventions: Other: read unfavorable article prior to answering questions
- Guideline favorable article (Active Comparator)
  Interventions: Other: read favorable article prior to answering questions

INTERVENTIONS:
Other: read unfavorable article prior to answering questions — article title: "Taking a hit on healthcare- why that's women's work"
  Other Names: Boston Globe, November 19, 2009; Section A17. Joan Vennochi.
  Arms: Guideline unfavorable article
Other: read favorable article prior to answering questions — read "A Backlash of Mistrust"
  Other Names: Washington Post; November 25, 2009. Ellen Goodman.
  Arms: Guideline favorable article

SUMMARY:
The purpose of this study was to determine attitudes regarding the 2009 USPSTF Guidelines for breast cancer screening for women in their 40's and assess the effect of one of two newspaper articles on their attitudes. The population studied was women seeing their private gynecologist for annual exams in the 39-49 year old age group.

DETAILED DESCRIPTION:
Subjects completed a baseline questionnaire listing demographics, previous experience with mammograms, and acquaintances with breast cancer. They then were randomly assigned one of two articles (one favorable and one unfavorable) that had been published in the newspaper regarding the USPSTF breast cancer screening guidelines. Their attitudes towards the safety of the guidelines and their willingness to comply with them was then measured.

ELIGIBILITY:
Inclusion Criteria:

* women aged 39-49 seeing their gynecologist for routine preventive care

Exclusion Criteria:

* women not aged 39-49
* women with breast cancer
* women not able to read English

Ages: 39 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 247 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Willingness to forgo mammograms from age 40-49 | within 15 minutes of completion of reading assigned article

SECONDARY OUTCOMES:
Do you feel that the mammogram recommendations safe? | within 15 minutes of completion of reading assigned article
Do attitudes regarding the breast cancer screening guidelines differ by acquaintance with breast cancer? | within 15 minutes of completion of reading assigned article
Does willingness to forgo mammograms in their 40's differ by previous "false alarms" with mammography? | within 15 minutes of completion of reading assigned article

CONTACTS AND LOCATIONS:
Overall Officials: Dale Magee, M.D., M.S., Principal Investigator — University of Massachusetts, Worcester; AuTumn Davidson, M.D., Study Director — University of Massachusetts, Worcester
Locations (4):
- United States (4):
  - UMassMemorial Medical Group- Auburn Gyn, Auburn, Massachusetts
  - Shrewsbury Ob-Gyn, Shrewsbury, Massachusetts
  - UMassMemorial Medical Group- OB-GYN, Shrewsbury, Massachusetts
  - Women's Health of Central Mass, Worcester, Massachusetts